CLINICAL TRIAL: NCT02541656
Title: Dynamic Preload Dependence Indices in Laparoscopic Surgery
Acronym: VPP Coelio
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2014-879
Record Dates: First submitted 2015-07-10; First posted 2015-09-04 (Estimated); Last update posted 2018-12-13 (Actual); Status verified 2018-12

CONDITIONS: Laparoscopic Surgery
Keywords: Preload dependence indices; pulse pressure variation; plethysmographic waveform of pulse oximetry variation; stroke volume variation; laparoscopy; pneumoperitoneum
MeSH Terms: conditions — Pneumoperitoneum | interventions — Laparoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- preloaddependence indice after volume expansion in laparoscopy (Experimental): The measurements of pulse pressure variation, plethysmographic waveform of pulse oximetry variation and stroke volume variation will be performed before pneumoperitoneum at the beginning of the surgery, and will be repeated after pneumoperitoneum insufflation applying each time modification of preload conditions (applying reverse Trendelenburg position followed by Trendelenburg position). The responses will be appreciated by the measurements of the stroke volume.
  Interventions: Procedure: Study of preload dependence indices after volume expansion in laparoscopy with Saldinger technique.

INTERVENTIONS:
Procedure: Study of preload dependence indices after volume expansion in laparoscopy with Saldinger technique. — The measurements of pulse pressure variation, plethysmographic waveform of pulse oximetry variation and stroke volume variation will be performed before pneumoperitoneum at the beginning of the surgery, and will be repeated after pneumoperitoneum insufflation applying each time modification of preload conditions (applying reverse Trendelenburg position followed by Trendelenburg position). The responses will be appreciated by the measurements of the stroke volume.

SUMMARY:
A goal-directed fluid management is definitely beneficial in high risk surgery. The fluid administration can be directed by cardiac output monitoring which evaluate the response to repeated fluid challenge or by preload dependence indices. These indices are not well validated in laparoscopic surgery while pneumoperitoneum can alter venous return or pulmonary compliance.

The aim of the study is to study the validity of pulse pressure variation to predict fluid response under laparoscopic conditions and to describe the effect of the pneumoperitoneum on the dynamic preload indicators, i.e. the pulse pressure variation, the plethysmographic waveform of pulse oximetry variation and the stroke volume variation.

ELIGIBILITY:
Inclusion Criteria:

* Need to laparoscopic colectomy or hepatic resection
* Written informed consent

Exclusion Criteria:

* Cardiac arrhythmia
* Esophageal and cervical pathologies
* Radial artery Allen test negative
* Allergy to anesthesic treatment, to egg or soja
* Severe kidney failure (estimated glomerular filtration rate < 30 ml/min)
* Age < 18 years old
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Assess the validity of pulse pressure variation (in %) | at Day 0
  Performing a fluid challenge after pneumoperitoneum insufflation, the association between pulse pressure variation value and stroke volume variation will be performed.
  Responder patients are defined by stroke volume augmentation > 15 %

SECONDARY OUTCOMES:
Threshold value to predict fluid response in laparoscopic conditions. | at Day 0
  A fluid challenge is performed after pneumoperitoneum insufflation to assess the fluid response and calculate the threshold value of fluid response.
Effect of the pneumoperitoneum insufflation on the preload dependence indices : plethysmographic waveform of pulse oximetry variation . | at Day 0
  The measures are performed after applying patient positioning which modify preload conditions. These measures are repeated before and after pneumoperitoneum insufflation and the values of each indices are compared.
Effect of the pneumoperitoneum insufflation on the preload dependence indices : stroke volume variation . | at Day 0
  The measures are performed after applying patient positioning which modify preload conditions. These measures are repeated before and after pneumoperitoneum insufflation and the values of each indices are compared.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon, Lyon, France